CLINICAL TRIAL: NCT07228364
Title: A Phase I Randomised, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD1613 Following Multiple Ascending Dose Administration in Participants With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Safety, Tolerability and Pharmacokinetics of AZD1613 in Adults With Autosomal Dominant Polycystic Kidney Disease
Acronym: PIONEER-PKD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9050C00002; Identifier Number (Registry Identifier: 174499)
Record Dates: First submitted 2025-10-23; First posted 2025-11-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: This is a Phase I, first-in-patient, randomized, single-blind, placebo-controlled study with a sequential MAD design in participants with autosomal dominant polycystic kidney disease (ADPKD). AZD1613 will be administered either subcutaneously or intravenously in up to 5 cohorts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be single-blinded in order to minimize bias in the collection and evaluation of data during its conduct.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - Cohort A1 (Experimental): Participants will receive 4 doses of AZD1613 or placebo on days 1, 29, 57 and 85.
  Interventions: Drug: AZD1613 - Part A; Drug: Placebo - Part A
- Part A - Cohort A2 (Experimental): Participants will receive 4 doses of AZD1613 or placebo on days 1, 29, 57 and 85.
  Interventions: Drug: AZD1613 - Part A; Drug: Placebo - Part A
- Part B - Chinese Cohort (Experimental): Participants will receive 4 doses of AZD1613 or placebo on days 1, 29, 57 and 85.
  Interventions: Drug: AZD1613 - Part A; Drug: AZD1613 - Part B; Drug: Placebo - Part B

INTERVENTIONS:
Drug: AZD1613 - Part A — Part A - Participants will be administered doses of AZD1613 on days 1, 29, 57, and 85 according to randomization in IRT.
Drug: Placebo - Part A — Part A - Participants will be administered doses of placebo on days 1, 29, 57, and 85 according to randomization in IRT.
  Arms: Part A - Cohort A1; Part A - Cohort A2
Drug: AZD1613 - Part B — Part B - Participants will be administered doses of AZD1613 on days 1, 29, 57, and 85 according to randomization in IRT.
  Arms: Part B - Chinese Cohort
Drug: Placebo - Part B — Part B - Participants will be administered doses of placebo on days 1, 29, 57, and 85 according to randomization in IRT.
  Arms: Part B - Chinese Cohort

SUMMARY:
A study to investigate safety, tolerability, and pharmacokinetics of AZD1613 following subcutaneous or intravenous administration in participants with autosomal dominant polycystic kidney disease (ADPKD).

DETAILED DESCRIPTION:
This Phase I, randomised, single-blind, placebo-controlled study will assess the safety and tolerability of AZD1613 and characterise the pharmacokinetics (PK) of AZD1613 in participants with autosomal dominant polycystic kidney disease (ADPKD), following subcutaneous (SC) or intravenous (IV) administration. Inclusion of participants receiving placebo is appropriate for benchmarking the safety and tolerability of AZD1613. Furthermore, the safety and PK profile will be evaluated in Chinese participants with ADPKD to assess any potential race effect in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADPKD Mayo Class (IB-IE), as per clinical diagnosis (MIC) assessed centrally. Genetic testing results will not be used for eligibility purposes
* eGFR = 45 to 90 mL/min /1.73m2
* Body weight ≥ 45 kg and body mass index within the range 18 to 35 kg/m2 (inclusive).
* Females are to be of non-childbearing potential

Exclusion Criteria:

* As judged by the investigator, any evidence of cardiac, vascular, and other renal conditions which in the investigator's opinion makes it undesirable for the participant to participate in the study.
* Positive hepatitis C antibody, hepatitis B virus surface antigen, or human immunodeficiency virus test, at screening.
* History of QT prolongation associated with other medications that required discontinuation of that medication.
* Congenital long QT syndrome.
* History of ventricular arrhythmia requiring treatment. Patients with atrial fibrillation/flutter and controlled ventricular rate HR < 100 bpm can be eligible as judged by the investigator.
* Haemoglobin below the lower limit of the normal range or any other clinically significant haematological abnormality as judged by the investigator.
* Any clinically important abnormalities in clinical chemistry, haematology, coagulation, or urinalysis results other than those specifically described as exclusion criteria herein, as judged by the investigator.
* Systolic BP > 160 mmHg or diastolic BP > 100mmHg or HR < 50 bpm or > 100 bpm at screening. Patients taking anti-hypertensive medication should be on a stable treatment regimen of antihypertensive therapy for at least 30 days prior to the screening visit.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, as considered by the investigator, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
* Kidney cyst interventions such as cyst aspiration or cyst fenestration within 12 weeks prior to screening and during the screening period, or such interventions planned or anticipated within the follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From randomization (Day 1) through end of follow-up (up to Day 189 ±3 days)
  Number of participants with at least one TEAE and SAE, including events leading to discontinuation or death; coded by system organ class and preferred term.
  Unit: participants.
Change From Baseline in Safety 12-Lead ECG QTcF | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in QT interval corrected using Fridericia's formula (QTcF) measured on single 12-lead safety ECGs.
  Unit: milliseconds (ms).
Change From Baseline in Safety 12-Lead ECG PR Interval | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in PR interval measured on single 12-lead safety ECGs.
  Unit: milliseconds (ms).
Change From Baseline in Safety 12-Lead ECG QRS Duration | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in QRS duration measured on single 12-lead safety ECGs.
  Unit: milliseconds (ms).
Change From Baseline in Heart Rate (12-Lead Safety ECG) | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in heart rate measured on single 12-lead safety ECGs.
  Unit: beats per minute (bpm).
Change From Baseline in ALT | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in alanine aminotransferase.
  Unit: U/L.
Change From Baseline in AST | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in aspartate aminotransferase.
  Unit: U/L.
Change From Baseline in Total Bilirubin | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in total bilirubin.
  Unit: mg/dL.
Change From Baseline in Serum Creatinine | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in serum creatinine.
  Unit: mg/dL.
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR; CKD-EPI 2021) | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in eGFR calculated using CKD-EPI 2021.
  Unit: mL/min/1.73 m².
Change From Baseline in INR | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in international normalized ratio- (INR).
  Unit: unitless.
Change From Baseline in Prothrombin Time (PT) | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in prothrombin time.
  Unit: seconds (s).
Change From Baseline in Activated Partial Thromboplastin Time (aPTT) | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in aPTT.
  Unit: seconds (s).
Change From Baseline in Urinary Albumin-to-Creatinine Ratio (UACR) | Baseline (Day -1) and scheduled visits through Day 189 ±3 days; UACR as triplicate first-morning voids per visit
  Change from baseline in UACR (geometric mean of triplicates at each visit).
  Unit: mg/g.
Change From Baseline in Systolic Blood Pressure | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in supine systolic blood pressure.
  Unit: mmHg.
Change From Baseline in Diastolic Blood Pressure | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in supine diastolic blood pressure.
  Unit: mmHg.
Change From Baseline in Heart Rate (Vital Signs) | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in supine heart rate.
  Unit: bpm.
Change From Baseline in Body Temperature | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in oral body temperature.
  Unit: °C.
Change From Baseline in Respiratory Rate | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in respiratory rate.
  Unit: breaths per minute.
Change From Baseline in Oxygen Saturation (SpO2) | Baseline (Day -1) and post-dose at scheduled visits through Day 189 ±3 days
  Change from baseline in pulse oximetry oxygen saturation.
  Unit: percent (%).

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of AZD1613 | Intensive PK sampling from Day 1 through Day 189 per protocol schedule
  Maximum observed serum concentration following subcutaneous or intravenous administration.
  Unit: µg/mL.
Area Under the Concentration-Time Curve to Last Quantifiable Concentration (AUClast) of AZD1613 | Intensive PK sampling from Day 1 through Day 189 per protocol schedule
  AUC from time zero to last quantifiable concentration.
  Unit: h·µg/mL (or day·µg/mL; align with bioanalytical report).
Area Under the Concentration-Time Curve From Time Zero to Infinity (AUCinf) of AZD1613 | Intensive PK sampling from Day 1 through Day 189 per protocol schedule
  AUC from time zero extrapolated to infinity.
  Unit: h·µg/mL (or day·µg/mL).
Area Under the Concentration-Time Curve Over the Dosing Interval at Steady State (AUCtau) of AZD1613 | Over the dosing interval (τ = 28 days) at steady state; sampling through Day 189
  AUC over the dosing interval at steady state.
  Unit: h·µg/mL (or day·µg/mL).
Time to Maximum Observed Serum Concentration (Tmax) of AZD1613 | Intensive PK sampling from Day 1 through Day 189 per protocol schedule
  Time to reach Cmax after dosing.
  Unit: hours (h).
Terminal Elimination Half-Life (t½) of AZD1613 | Intensive PK sampling from Day 1 through Day 189 per protocol schedule
  Half-life associated with terminal slope (λz) of the concentration-time curve.
  Unit: hours (h) or days (d).
Incidence of Anti-Drug Antibodies (ADA) to AZD1613 | Predose on dosing days and during follow-up through Day 189 ±3 days
  Number of participants with ADA-positive response based on validated tiered assay (screen and confirm).
  Unit: participants.
ADA Titer to AZD1613 | Predose on dosing days and during follow-up through Day 189 ±3 days
  Titer among confirmed ADA-positive samples.
  Unit: reciprocal dilution (titer).
Change From Baseline in PD Markers of PAPPA-1 Inhibition | Baseline to scheduled post-dose time points through Day 189 ±3 days
  Change from baseline in pharmacodynamic marker of PAPPA-1 inhibition.
  Unit: ng/mL (or assay-specific unit).

CONTACTS AND LOCATIONS:
Locations (15):
- United States (8):
  - Research Site, Birmingham, Alabama
  - Research Site, Loma Linda, California
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Lenexa, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, San Antonio, Texas
- China (6):
  - Research Site, Chengdu
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Xiamen
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/